CLINICAL TRIAL: NCT00620243
Title: Pilot Study to Evaluate 18F-fluorodeoxyglucose (FDG) Positron Emission Tomography /Computed Tomography (PET/CT) in Prediction of Early Response to Chemotherapy in Ovarian Cancer.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 04-064
Record Dates: First submitted 2008-01-25; First posted 2008-02-21 (Estimated); Last update posted 2012-01-09 (Estimated); Status verified 2012-01

CONDITIONS: Ovarian Cancer
Keywords: Ovarian cancer; PET; CT; 04-064
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): The study will evaluate the potential of PET imaging to identify early responders to chemotherapy. Patients entered into this study will undergo FDG PET within 2 weeks prior to chemotherapy and prior to initiation of the second course of chemotherapy. All images will be carried out in the same manner with respect to equipment, acquisition parameters, and time post injection, to ensure that changes in standard uptake value(SUV) correlate with metabolic changes. This will be correlated with response determined by changes in serum CA 125 levels.
  Interventions: Procedure: 1: FDG PET

INTERVENTIONS:
Procedure: 1: FDG PET — The study will evaluate the potential of PET imaging to identify early responders to chemotherapy. Patients entered into this study will undergo FDG PET within 2 weeks prior to chemotherapy and prior to initiation of the second course of chemotherapy. All images will be carried out in the same manner with respect to equipment, acquisition parameters, and time post injection, to ensure that changes in standard uptake value(SUV) correlate with metabolic changes. This will be correlated with response determined by changes in serum CA 125 levels.

SUMMARY:
We hypothesize that 18FDG Positron Emission Tomography (FDG PET) imaging, carried out after the first cycle of chemotherapy, will identify responders, thus permitting early termination of potential toxic therapy in non- responders leading to a significant decrease in morbidity and cost. The value of PET imaging as an early predictor of response to chemotherapy has been shown in other cancers.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven ovarian cancer at diagnosis of any stage.
* Patients with evidence of disease that is radiographically measurable (CT scan)
* Patients have planned to undergo standard chemotherapy. Dose and schedule will be determined per treating physician

Exclusion Criteria:

* Patients with any other malignancy active within 5 years except for non-melanoma skin cancer, or carcinoma in situ of the cervix.
* Patients with an active infection
* Patients of childbearing potential are excluded from this study.
* Patients who have expected survival < 3 months.
* Patients not planning or able to receive the outlined chemotherapy regimen as part of standard practice.
* Patient unable to complete study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2004-06; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Partial metabolic response (PMR) - A reduction of a minimum of 15-25% in tumour 18FDG SUV after one cycle of chemotherapy, and greater than 25% after more than one treatment cycle. | Conclusion of the study
Partial metabolic response (PMR) - A reduction of a minimum of 15-25% in tumour 18FDG SUV after one cycle of chemotherapy, and greater than 25% after more than one treatment cycle. | Completion of study
Complete metabolic response (CMR) - Complete resolution of 18FDG uptake within the tumour volume so that it was indistinguishable from surrounding normal tissue. | completion of study
Progressive metabolic disease- increase in 18FDG tumour SUV of greater than 25% within tumour region defined on the baseline scan, visible increase in the extent of 18FDG tumour uptake (>20% in the longest dimension). | completion of study
Stable metabolic disease (SMD) -An increase in tumour 18FDG SUV of less than 25% or a decrease of less than 15% and no visible increase in extent of 18FDG uptake in tumor (>20% in the longest dimension). | completion of study

CONTACTS AND LOCATIONS:
Overall Officials: Neeta Pandit-Taskar, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Related Info — http://www.mskcc.org